CLINICAL TRIAL: NCT04829669
Title: Prospective Study to Assess, Outcomes and Healthcare Resource Use of Current Standard of Care for Patients With Moderate or sEvere MDD Requiring Urgent Symptom Control in a Psychiatric Emergency: POWER
Brief Title: A Study of Participants With Moderate or Severe Major Depressive Disorder (MDD) Requiring Urgent Symptom Control in a Psychiatric Emergency
Acronym: POWER
Status: Withdrawn | Type: Observational
Why Stopped: The study has faced delays in past years - COVID-19 pandemic and recruitment of a sensitive population. New challenges have led to this cancellation decision.
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109009; 54135419MDD4003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Major Depressive Disorder (MDD) and Active Suicidal Ideation with Intent: Participants with MDD (moderate or severe) and active suicidal ideation with intent as defined/confirmed by healthcare team will be enrolled and treated in accordance with routine clinical practice. The primary data source for this study will be the medical chart review, carer and clinician-reported outcome measures records of each participant.

SUMMARY:
The purpose of the study is to describe the clinical outcomes (severity of depression, severity of suicidality & frequency of suicidal thinking, suicide events) and quality of life (QoL) of participants with symptoms of major depressive disorder (MDD) that have current suicidal ideation with intent.

ELIGIBILITY:
Inclusion Criteria:

For Participant and Carer

* Capacity to provide consent
* Must sign an informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements
* Sufficient command of English language to understand the study information and requirements For Participant
* Participant must be deemed to have current suicidal ideation with intent at the point of study enrollment and be within four days of presenting with suicidal ideation with intent in relation to the current episode For Carer
* Participant and/ or carer report that the carer has a personal relationship with the patient and provides unpaid support or care

Exclusion Criteria:

* Capacity to provide consent
* Participant is known to be diagnosed with any of the following conditions: mania, bipolar disorder, psychotic disorder, depression with psychotic features, autism, dementia, intellectual disability
* Participant is known to be diagnosed with any of the following conditions: mania, bipolar disorder, psychotic disorder, depression with psychotic features, autism, dementia, intellectual disability

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population consists of participants with confirmed Major Depressive Disorder (MDD) and active suicidal ideation with intent as per healthcare team opinion.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Severity of Depression as Assessed by the Montgomery-asberg Depression Rating Scale (MADRS) | Baseline, up to 90 days
  MADRS is a clinician-rated scale designed to measure changes in depression severity due to antidepressant treatment. The MADRS consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms) for a total possible score of 60. Higher scores represent a more severe condition. The Structured Interview Guide for the MADRS (SIGMA) will be used for the administration of the MADRS assessment.
Change From Baseline in Severity of Suicidality as Assessed by Clinical Global Impression-Severity of Suicidality Revised (CGI-SS-R) Score | Baseline, up to 90 days
  CGI-SS-R is derived from the Clinical Global Impression Severity Scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participant's illness. The CGI-SS-R rating is scored on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants). A higher score indicates a more severe condition and a reduction in score indicates improvement (that is, lower severity of suicidality).
Change From Baseline in Suicide Ideation and Behavior Assessment Tool (SIBAT) Module 7 (Clinician-rated Frequency of Suicidal Thinking [FoST]) Score | Baseline, up to 90 days
  SIBAT is assessment tool that captures suicidal ideation, behavior, and risk. It permits assessment of change in suicidal ideation and behavior and documents clinician assessment of severity of suicidality and suicide risk. SIBAT has 8 modules divided into 2 major divisions: patient-reported section (Modules 1-5) and clinician-rated section (Modules 6-8). Clinician-rated section has modules for semi-structured interview, clinical global impressions of current severity of suicidality and imminent suicide risk, clinical global impression of long-term suicide risk, and clinical judgment of optimal suicide management. The score anchor point as in participant report frequency of suicidal thinking that is, response options from never to all the time. Module 7-FoST score ranges from 0-5; higher score indicates more severe condition. Negative change in score indicates improvement.
Change From Baseline in European Quality of Life (EuroQol) 5-Dimension 5-Level Questionnaire (EQ-5D-5L) Scores | Baseline, up to 90 days
  The EQ-5D-5L is a generic measure of health status. It is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).

SECONDARY OUTCOMES:
Number of Participants with Inpatient and Outpatient Care Across Specific Settings and Consultation With Different Healthcare Professionals (HCPs) | Up to 90 days
  Number of participants with Inpatient and outpatient care across specific settings and consultation with different healthcare professionals (HCPs) will be reported.
Number of Resources Used to Reduce the Risk for Suicide | Up to 90 days
  Number of Resources (hospitalization, close surveillance, crisis team support etc.) used to reduce the risk for suicide will be reported.
Number of Participants who Used Psychopharmacological and Non-pharmacological Drug Therapies | Up to 90 days
  Number of participants who psychopharmacological drug therapies and non-pharmacological therapies including psychological therapies and electroconvulsive therapy will be reported.
Care Burden as Assessed by EQ-5D-5L Score | Up to 90 days
  The EQ-5D-5L is a generic measure of health status. It is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Care Burden as Assessed Work productivity and Activity Impairment Questionnaire (WPAI) Score | Up to 90 days
  The WPAI consist of four types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. Outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity that is worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.